CLINICAL TRIAL: NCT01923818
Title: Randomized,Double-blind Trial Comparing the Effects of a Rivaroxaban Regimen During the First 30 Days,Versus Aspirin for the Acute Treatment of TIA or Minor Stroke
Brief Title: Treatment of Rivaroxaban Versus Aspirin for Non-disabling Cerebrovascular Events
Acronym: TRACE
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Xijing-TRACE
Record Dates: First submitted 2013-07-19; First posted 2013-08-16 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Ischemic Stroke; TIA
Keywords: rivaroxaban; aspirin; new oral anticoagulant; TIA; acute minor ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- aspirin (Active Comparator): Receiving a 100-mg dose of aspirin and placebo rivaroxaban from day 1 to day 30
  Interventions: Drug: Aspirin; Drug: placebo
- Rivaroxaban 5mg (Experimental): Receiving a 5-mg dose of rivaroxaban and placebo aspirin from day 1 to day 30
  Interventions: Drug: rivaroxaban; Drug: placebo
- rivaroxaban 10mg (Experimental): Receiving a 10-mg dose of rivaroxaban and placebo aspirin from day 1 to day 30
  Interventions: Drug: rivaroxaban; Drug: placebo

INTERVENTIONS:
Drug: rivaroxaban — orally active direct factor Xa inhibitor
  Other Names: BAY 59-7939; Xarelto
  Arms: Rivaroxaban 5mg; rivaroxaban 10mg
Drug: Aspirin — non-steroidal anti-inflammatory drugs
  Other Names: Acetylsalicylic acid
  Arms: aspirin
Drug: placebo

SUMMARY:
Transient ischemic attack (TIA) or minor ischemic stroke has a high risk of early recurrent stroke. As the golden standard, aspirin effect modestly on acute ischemic stroke, and slightly increase the risk of intracerebral hemorrhage. Recently, rivaroxaban, a new oral anticoagulant, is proved to be as effective as traditional anticoagulants, while carrying significantly less risk of intracranial hemorrhage.

The TRACE trial is a randomized, double-blind, multicenter, controlled clinical trial in China. The investigators will assess the hypothesis that a 30-days rivaroxaban regimen is superior to aspirin alone for the treatment of high-risk patients with acute nondisabling cerebrovascular event.

DETAILED DESCRIPTION:
The TRACE study is a randomized, double-blind clinical trial with a target enrollment of 3,700 Chinese patients. Two subtypes of patients will be enrolled: I, acute disabling ischemic stroke (<24 hours of symptoms onset); II, acute TIA (<24 hours of symptoms onset).

Patients will be randomized into 3 groups:

* Receiving a 100-mg dose of aspirin and placebo rivaroxaban from day 1 to day 30
* Receiving a 5-mg dose of rivaroxaban and placebo aspirin from day 1 to day 30
* Receiving a 10-mg dose of rivaroxaban and placebo aspirin from day 1 to day 30

The primary efficacy end point is percentage of patients with new stroke (ischemic or hemorrhage) at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (male or female ≥18 years old)
* Acute nondisabling ischemic stroke (NIHSS ≤3 at the time of randomization) that can be treated with study drug within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* TIA (neurologic deficit attributed to focal brain ischemia, with resolution of the deficit within 24 hours of symptom onset), that can be treated with investigational medication within 24 hours of symptoms onset. Symptom onset is defined by the "last see normal" principle
* Informed consent signed

Exclusion Criteria:

* Diagnosis of hemorrhage or other pathology, such as vascular malformation, tumor, abscess or other major nonischemic brain disease, on baseline head CT or MRI scan
* mRS score >2 at randomization (premorbid historical assessment)
* NIHSS ≥4 at randomization
* Clear indication for anticoagulation (atrial fibrillation, mechanical cardiac valves, deep venous thrombosis, pulmonary embolism or known hypercoagulable state)
* Contraindication to investigational medications
* Thrombolysis for ischemic stroke within preceding 7 days
* History of intracranial hemorrhage
* Current treatment (last dose given within 10 days before randomization) with heparin therapy or oral anticoagulation
* Gastrointestinal bleed or major surgery within 3 months
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
* TIA or minor stroke induced by angiography or surgery
* Severe noncardiovascular comorbidity with life expectancy <3 months
* Women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test result
* Severe renal failure, defined as Glomerular Filtration Rate (GFR) <30 ml/min Severe hepatic insufficiency (Child-Pugh score B to C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3700 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with new stroke (ischemic or hemorrhage) | 90 days

SECONDARY OUTCOMES:
Percentage of patients with new clinical vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) | 30 days
mRS score changes (continuous) and dichotomized at percentage with score 0 to 2 versus 3 to 6 | 30 days and 90 days
Changes in NIHSS scores | 90 days
moderate to severe bleeding events | 90 days
Total mortality | 90 days
Adverse events/severe adverse events reported by the investigators | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gang Zhao, M.D., Principal Investigator — Neurology Department,Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Yang F, Jiang W, Bai Y, Han J, Liu X, Zhang G, Zhao G. Treatment of Rivaroxaban versus Aspirin for Non-disabling Cerebrovascular Events (TRACE): study protocol for a randomized controlled trial. BMC Neurol. 2015 Oct 12;15:195. doi: 10.1186/s12883-015-0453-7. PMID 26458895